CLINICAL TRIAL: NCT05642416
Title: Intermittent Bolus Versus Continuous Infusion Erector Spinae Catheters for Median Sternotomy Incisions: A Prospective Randomized Controlled Trial
Brief Title: Intermittent Bolus vs Continuous Infusion Via ESP Catheters RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Avanos Medical (Other)
Responsible Party: Principal Investigator, Patrick Forrest, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15737
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two treatment groups (one with continuous infusion of drug and the other with bolus via ESP catheter)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only people who will know the treatment arm that has been assigned to the participant are the research coordinator who randomized them and the regional anesthesia team. The patient, nursing team, and research coordinator performing outcomes assessments will all be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continuous Infusion (Active Comparator): Will receive a continuous infusion of pain medication (0.2% ropivacaine at a rate of 10mL per hour- 5mL per side per hour) via erector spinae plane (ESP) catheter for their postoperative pain following median sternotomy incision.
  Interventions: Drug: Continuous Infusion of ropivacaine
- Intermittent Bolus (Experimental): Will receive intermittent boluses of pain medication (30mL bolus of 0.2% ropivacaine every three hours) via erector spinae plane (ESP) catheter for their postoperative pain following median sternotomy incision.
  Interventions: Drug: Intermittent bolus of ropivacaine

INTERVENTIONS:
Drug: Continuous Infusion of ropivacaine — Continuous infusion of ropivacaine
  Arms: Continuous Infusion
Drug: Intermittent bolus of ropivacaine — Intermittent bolus of ropivacaine
  Arms: Intermittent Bolus

SUMMARY:
The purpose of this prospective randomized controlled trial is to compare the effectiveness of two different delivery methods for postoperative pain management following cardiac surgery requiring median sternotomy: intermittent programmed LA bolus versus continuous LA infusion through ESP catheters. Effectiveness of analgesia will be assessed based on the subjects' NRS pain scores and opioid consumption. The primary outcome measure will be the patients' opioid consumption over the course of the 72 hours following surgery. Secondary outcomes measures that will be evaluated include NRS pain scores, intensive care unit (ICU) length of stay, and time to first dose of antiemetic in the postoperative period. It is hypothesized that the use of intermittent programmed LA boluses will provide better analgesia compared to continuous LA infusion through ESP catheters. The findings of this study will provide guidance regarding the optimal method of delivery for postoperative pain management in patients following cardiac surgery.

DETAILED DESCRIPTION:
The purpose of this prospective randomized controlled trial is to compare the effectiveness of two different delivery methods for postoperative pain management following cardiac surgery requiring median sternotomy: intermittent programmed LA bolus versus continuous LA infusion through ESP catheters. Effectiveness of analgesia will be assessed based on the subjects' NRS pain scores and opioid consumption. The primary outcome measure will be the patients' opioid consumption over the course of the 72 hours following surgery. Secondary outcomes measures that will be evaluated include NRS pain scores, intensive care unit (ICU) length of stay, and time to first dose of antiemetic in the postoperative period. It is hypothesized that the use of intermittent programmed LA boluses will provide better analgesia compared to continuous LA infusion through ESP catheters. The findings of this study will provide guidance regarding the optimal method of delivery for postoperative pain management in patients following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent elective cardiac surgery requiring median sternotomy for surgical exposure (i.e. CABG, aortic/mitral/tricuspid valve replacements) receiving ESP catheter preoperatively
* Age 18-90

Exclusion Criteria:

* Placement and/or existence of cardiac assist devices (LVAD, RVAD, Balloon Pump, Impella)
* Neurocognitive dysfunction
* Patients who expire before extubation
* Non-English speaking
* Daily opioid therapy prior to surgery
* History of substance abuse
* BMI > 45

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours post-op
  Opioid consumption (MME) over the course of the 72 hours following surgery

SECONDARY OUTCOMES:
NRS Pain Scores (10) | 72 post-op
  Numeric rating scale for pain (rated 0=no pain through 10= worst imaginable pain)
ICU length of stay | 72 hours post-op
  Time from post-op to step-down from ICU
Quality of Recovery 15 (QoR-15) score | 72 hours post-op
  Quality of Recovery 15 (QoR-15) score: 15 question survey (0=very poor recovery through 150=excellent recovery)
Time to first antiemetic | 72 hours post-op
  Time to first antiemetic

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data available to other researchers.